CLINICAL TRIAL: NCT00338078
Title: Nocturnal Oxygen Treatment in Heart Failure and Cheyne-Stokes Respiration. A Randomized Double-Blind Placebo Controlled Cross-Over Study
Brief Title: Nocturnal Oxygen Treatment in Heart Failure and Cheyne-Stokes Respiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 241/98, dnr 98-165
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Device: nocturnal oxygen treatment from oxygen concentrators

SUMMARY:
The purpose of this study is to determine whether oxygen therapy during sleep improves quality of life, exercise capacity and heart function among patients with chronic heart failure and central sleep apnea.

DETAILED DESCRIPTION:
Oxygen therapy reduces the number of central apneas among patients with congestive heart failure but it is unknown whether quality of life and heart function also improve. We aim to test whether the quality of life, exercise capacity and heart function are improved with nocturnal oxygen therapy during 6 weeks with nocturnal oxygen from oxygen concentrator or nocturnal air from placebo concentrator.

ELIGIBILITY:
Inclusion Criteria:

* Stable heart failure with left ventricular dysfunction
* Cheyne-Stokes respiration with central AHI>15 and obstructive AHI<5

Exclusion Criteria:

* Heart infarction within 3 months.
* Dementia
* Chronic obstructive pulmonary disease and daytime hypoxemia.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 1999-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Exercise capacity
Quality of life (SF-36, Minnesota, Living with heart failure questionnaire)
Brain natriuretic peptide (BNP)

SECONDARY OUTCOMES:
Echocardiography
Radionuclide determination of ejection fraction
Mortality and hospitalization for cardiovascular causes (combined and individually)
Hospitality anxiety and depression scale
Epworth sleepiness scale
Karolinska sleepiness scale
Routine lab (haemoglobins, thyroid status, creatinin)
Urinary catecholamines
Urinary cortisol
Polysomnography
Arrhythmias from 24 hour Holter-ECG registration
Heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, PhD, Principal Investigator — Dept Respiratory Medicine, University Hospital, Umeå
Locations (1):
- Dept of respiratory medicine, Umeå, Sweden